CLINICAL TRIAL: NCT05767177
Title: Small Intestinal Ketogenesis - Potential Significance for Type 2 Diabetes in Obesity
Brief Title: Jejunal Ketogenesis and Type 2 Diabetes
Acronym: But2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Ketogen05
Record Dates: First submitted 2023-02-16; First posted 2023-03-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Morbid; Diabetes Mellitus, Type 2; Intestines; Incretins
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Carbohydrate Diet vs High Fat Diet (Experimental): In the current project, the situation applies to individuals with obesity (body mass index (BMI) 35 to 45 kg/m2). In one case the diet is of the type "high-carbohydrate diet" and in the other case "high-fat diet". The idea is that the research subjects should subsist on these diets for the respective 14 days. The energy content of the diet periods must be the same and correspond to the participants' daily needs. Each participant is drawn to one diet for 2 weeks. After a break of at least 3 weeks, the second diet is taken for 2 weeks.
  Interventions: Other: Glucemia following Mixed Meal Test; Other: Enteroscopy - mucosal ketogenic activity as well as glucose transport

INTERVENTIONS:
Other: Glucemia following Mixed Meal Test — On day 12 of each diet, a venous catheter is placed in one arm for blood sampling and the research person must answer questions about any gastrointestinal complaints in connection with the current diet. At approximately 09:00, the research subject may eat a brunch for approximately 15 minutes (sandwich, juice, fried egg and sausage; 550-600kcal). Venous blood samples are taken before and 15, 30, 45, 60, 90 and 120 minutes after the meal.
Other: Enteroscopy - mucosal ketogenic activity as well as glucose transport — On day 14 of each diet period, an enteroscopy is performed. This step is performed to obtain samples (biopsy) of the mucosa of the small intestine (duodenum and jejunum) and is performed at the Gastro-endoscopic departments SU-Sahlgrenska, or SU-Eastern hospital. Endoscopy is experienced by some individuals as unpleasant, which is why local anesthesia and sometimes sedation (midazolam + pethidine or rapifen) can be offered according to standard routine in the endoscopy department.

SUMMARY:
The goal of this cross-over study in obese subjects is to learn about the common co-morbidity type 2 diabetes and the local formation of ketone bodies. The type of study is an exploratory trial with the participants as own controls. The main questions it aims to answer are: 1. Does food intake-induced ketogenesis exist in the small intestine of obese individuals? 2. Are insulin resistance, the incretin GLP-1 release and the glucose transporter SGLT1 affected in obese individuals without type 2 diabetes in the same way as those with type 2 diabetes?

DETAILED DESCRIPTION:
The investigators have recently shown that the mucosa in the middle small intestine, the jejunum, in human volunteers produce ketones bodies.This situation is thus contrary to the common view that ketone bodies are formed by the liver during fasting/starvation. Obesity is commonly associated with hyperglycaemic conditions and diabetes mellitus type 2.This has given rise to the question of whether obesity results in disturbances in the intestinal food-induced ketogenesis and whether this influence contributes to the development of type 2 diabetes mellitus?

The project's questions are therefore:

1. Does food intake-induced ketogenesis exist in the small intestine of obese individuals?
2. Are insulin resistance, the incretin GLP-1 release and the glucose transporter SGLT1 affected in obese individuals without type 2 diabetes in the same way as those with type 2 diabetes?
3. If no to 2: What is the difference?

ELIGIBILITY:
Inclusion Criteria:

* BMI 35 to 45 kg/m2

Exclusion Criteria:

* Insulin-treated diabetes
* Sequelae of previous diabetes-associated disease (foot, eyes and kidneys, or cardiovascular incident, etc.)
* Diabetes, hypertension, lipid disorder that has not been stabilized for at least 1 month by adequate pharmacological treatment
* Continuous NSAID use
* Preferably otherwise medication-free (exceptions can be made)
* Not operated on in the abdomen (appendectomy excluded)
* Previously known organic gastrointestinal disease, except for gastroesophageal reflux disease (GERD)
* Smokers
* Pregnancy and breastfeeding
* History of drug abuse or other circumstances deemed to jeopardize the patient's ability to participate in the research project

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Glucemia following a Mixed Meal Test: | On day 12 of the respective diet
  The study participant arrives fasted and a venous catheter is placed in one arm for blood sampling. The research subject may eat a brunch for approximately 15 minutes (sandwich, juice, fried egg and sausage; 550-600kcal) and the p-glucose (mM) is checked at 120 min.
  The glucemia after the test meal will be compared in high-carbohydrate diet and high-fad diet (paired samples).

SECONDARY OUTCOMES:
Enteroscopy: ketogenic activity in the small intestine | On day 14 of the respective diet
  The biopsy material is fixed deep-frozen for later analyses.The ketonic activity is represented by the activity the ketogenic enzyme mitochondrial 3-hydroxy-3-methylglutaryl-CoA synthase (HMGCS2) in the tissue.
  Immunofluorescence of antibodies (giving the geography in the duodenal/jejunal mucosa) and western blotting (semi-assessment compared to a steadily-expressed factor in the mucosa, glyceraldehyde 3-phosphate dehydrogenase (GAPDH). The HMGCS2 will be given as ratio to GAPDH. The western blots in the high-carbohydrate diet will be compared to high-fad diet in each individual (paired samples).
Enteroscopy: mucosal glucose-transport capacity | On day 14 of the respective diet
  A part of the biopsy-material is kept a short time (<2h) in oxygenated preservation medium. The biopsies are then mounted in Ussing chambers for in-vitro functional studies. Activity of the sodium-glucose linked transporter 1 (SGLT1) is measured as the electrogenic response of 10 mM D-glucose, Iep (µA/mm2), given to the luminal compartment of the Ussing chamber. The net change is the % change of Iep from baseline in the glucose-free condition, to Iep after the addition of glucose to a concentration of 10%. The net change after the high-carbohydrate diet will be compared to the one after high-fat diet in each individual (paired samples).

OTHER OUTCOMES:
Glucemia, insulinemia and GLPi-emia following the Mixed Meal Test | On day 12 of the respective diet
  The study participant arrives fasted and a venous catheter is placed in one arm for blood sampling. The research subject may eat a brunch for approximately 15 minutes (Mixed Meal Test (MMT): sandwich, juice, fried egg and sausage; 550-600kcal) and the p-glucose (mM), p-insulin (µUnits/mL) and p-GLP1 (pM) is checked after 15, 30, 45, 60, 90 and120 min.
  The aggregated responses to MMT (linear area under the curve minus the baseline value) over 120 min of the respective agent are compared in high-carbohydrate diet and high-fad diet.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fändriks, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Dept of Surgery, Sahlgrenska Universityhospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
This is an exploratory studie with a rather small number of participants.

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT05767177/Prot_002.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT05767177/ICF_003.pdf